CLINICAL TRIAL: NCT06759584
Title: Continuous Versus Pulsed Dexamethasone Phonophoresis in Management of TMD. A Comparative Clinical Study
Brief Title: Management of Temporomandibular Disorders (TMD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Tarek Abdelbarry, Lecturer of Oral and Maxillofacial Surgery, Minia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Temporomandibular disorders
Record Dates: First submitted 2024-12-28; First posted 2025-01-06 (Actual); Last update posted 2025-01-06 (Actual); Status verified 2023-04

CONDITIONS: Temporomandibular Disorder
MeSH Terms: conditions — Temporomandibular Joint Disorders | interventions — Dexamethasone; Phonophoresis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group A (Active Comparator): About 20 patients who will receive dexamethasone gel and continuous phonophoresis
  Interventions: Drug: Dexamethasone
- Group B (Active Comparator): About 20 patients who will receive dexamethasone and pulsed phonophoresis
  Interventions: Drug: Dexamethasone
- Group C (Active Comparator): About 20 patients who will receive acoustic gel and continuous phonophoresis
  Interventions: Drug: Dexamethasone
- Group D (Active Comparator): About 20 patients who will receive acoustic gel and pulsed phonophoresis
  Interventions: Drug: Dexamethasone

INTERVENTIONS:
Drug: Dexamethasone — To Compare clinical outcome of dexamethasone phonophoresis in a (continuous and pulsed) maneuver for management of Temporomandibular Disorders
  Other Names: Phonophoresis

SUMMARY:
Temporomandibular disorders (TMD) are a group of pathologies of the temporomandibular joint, their muscles, and related structures. It is considered a musculoskeletal disorder of the masticatory system, and it has a 25% prevalence in overall population.

In 3% - 7% of the population, pain and dysfunction leads to the need for treatment . The etiology of TMD is multifactorial .

DETAILED DESCRIPTION:
Temporomandibular disorder is characterized by signs and symptoms that include pain, muscle tenderness, joint noises, and a limited range of motion.

The normal distance of mouth opening (inter-incisal distance) is 53 - 58mm. A minimal limit of 40 mm might be used to identify patients with limited aperture, whereas 35 mm is the necessary criteria for diagnosing disc displacement without reduction after unforced maximal aperture .

Due to all symptoms involved, a multidisciplinary approach is recommended for effective management of such cases. Conservative management of TMD treatment includes occlusal splints; physical therapy; oral medication (NSAIDs and muscle relaxants); and orthodontic treatment. Physical therapy is an important option used to reduce pain and inflammation and to improve oral mobility and function.

Phonophoresis is a method which intensifies the delivery of a topical agent into underlying tissues by ultrasound . It has been used with topical application of steroids, salicylate, anesthetic agents, methly nicotinate, NSAID . It is one of the many modalities for the treatment of musculoskeletal disorders.

Corticosteroids are used to reduce inflammation in systemic disease, local tendanitis, myositis, and other soft tissues. While these drugs are most often taken orally, they have also been applied transcutaneously by rubbing, injection, electrical current, or ultrasound. Transcutaneous drug delivery has a faster distribution rate into the system once it diffuses through the outer layer of the skin, quickly reaching the arterioles in the epithelium it is carried out systemically. As the blood moves through the vessels, part of the drug leaks into the surrounding tissues. These advantages have justified researching different methods to enhance transcutaneous delivery, avoiding unnecessary prolonged drug contact.

ELIGIBILITY:
Inclusion Criteria:

* patients 20- 50 years showing TMD
* pain > 3 on Visual Analog scale (VAS)
* failed pharmacological treatment

Exclusion Criteria:

* electrical stimulator or pacemaker
* cancer or any other severe or mental diseases
* osteoarthritis, inflammation, infection, or radiation on the TMJ articulation,
* joint cement or plastic components on TMJ articulation

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2023-04-28 (Actual); Primary Completion 2024-02-20 (Actual); Study Completion 2024-02-28 (Actual)

PRIMARY OUTCOMES:
Management of Pain | First 24 hours after The Operations
  Pain scores will be recorded on visual analog scale (VAS) using a 0 to 10 pain score basis with 0 being no pain and 10 being the worst pain the patient had ever experienced.

CONTACTS AND LOCATIONS:
Overall Officials: Tarek Abdelbarry, Lecturer, Principal Investigator — Faculty of Dentistry, Minia University
Locations (1):
- Faculty of Dentistry, Minia University, Minya, Egypt

IPD SHARING:
Plan to Share IPD: Undecided